CLINICAL TRIAL: NCT06545851
Title: Automatic Oxygen Titration Versus Constant Oxygen Flow Rates During Exercise Training in Hypoxemic People With Chronic Lung Disease - a Randomized, Double-blind, Controlled Cross-over Pilot Study
Brief Title: Effects of an Automatic Oxygen Titration System in People With Hypoxemia During Exercise Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Principal Investigator, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: O2matic exercise training
Record Dates: First submitted 2023-08-08; First posted 2024-08-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hypoxaemia; Chronic Lung Disease
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participant and investigator is blinded to the type of oxygen supply (constant flow or automatic titrating flow).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excercise Training Order A and B (Experimental): The first series of five exercise trainings (A) involves supplemental oxygen therapy, with automatically titrated oxygen flow rates to maintain an oxygen saturation of 90-94% (A). The second series of five exercise trainings employs supplemental oxygen therapy with constant flow rates (B), as prescribed.
  Interventions: Other: Oxygen therapy - constant oxygen flow; Other: Oxygen therapy - automatic titrating oxygen flow
- Excercise Training Order B and A (Experimental): The first series of five exercise trainings employs supplemental oxygen therapy with constant flow rates (B), as prescribed.The second five series of five exercise trainings involves supplemental oxygen therapy, with automatically titrated oxygen flow rates to maintain an oxygen saturation of 90-94% (A).
  Interventions: Other: Oxygen therapy - constant oxygen flow; Other: Oxygen therapy - automatic titrating oxygen flow

INTERVENTIONS:
Other: Oxygen therapy - constant oxygen flow — During five exercise training sessions, oxygen therapy is delivered via prescribed constant oxygen flow
Other: Oxygen therapy - automatic titrating oxygen flow — During five exercise sessions, oxygen therapy is delivered via an automatically titrated oxygen flow rate to maintain an SpO2 target of 90-94%.

SUMMARY:
Long-term oxygen therapy is a fundamental treatment modality for patients with chronic hypoxaemic lung disease. Typically, oxygen is administered at a constant flow rate. However, due to fluctuating activity levels, patients' oxygenation status can vary, potentially leading to oxygen desaturation and increased dyspnoea.

Emerging evidence suggests that automatic oxygen titration - a method of adjusting oxygen flow in response to current oxygen saturation - may have acute advantages over constant oxygen flow.

The primary objective of this study is to investigate the effect of automatic oxygen titration compared to prescribed constant oxygen flow rates on patients' perceived dyspnoea during exercise endurance training.

DETAILED DESCRIPTION:
Rationale:

Hypoxaemia is common in people with chronic lung disease and can affect exercise tolerance. Oxygen therapy is then recommended.

Oxygen supplementation is usually delivered at constant oxygen flow rates. Only a few studies have investigated the short-term effects of automated oxygen delivery compared to a constant oxygen flow rate during exercise tests (e.g. 6-minute walk test, shuttle walk tests). These studies have shown that automatic oxygen delivery can lead to an acute increase in exercise capacity, including an improvement in the perception of breathlessness. The use of automated oxygen delivery during endurance exercise has not been studied. The most common reason for stopping prolonged exercise in patients with chronic lung disease is dyspnoea. Therefore, the use of automatic oxygen delivery in a pulmonary rehabilitation clinic could be beneficial in the context of personalised therapy for patients requiring oxygen if it further reduces dyspnoea, potentially enabling the patient to train their endurance even better.

Therefore, the primary aim of this study was to investigate whether the use of automatic oxygen supplementation versus constant oxygen supplementation has a different effect on the perception of dyspnoea in patients with hypoxaemia during endurance exercise.

Design:

This study is designed as a randomised, double-blind, controlled cross-over trial. Participants will first undergo a cycle-based peak work rate test to determine their individual maximal peak work rate. They then take part in two sets of five endurance training sessions. One set is performed with a constant oxygen flow prescribed for each participant, while the other uses automatic oxygen titration. The order in which these two sessions are performed is randomised.

ELIGIBILITY:
Inclusion Criteria:

* Chronic lung disease
* Hypoxemia (pO2< 55mmHg) under room air conditions (rest or during exercise) or SpO2<88% during exercise
* established Long-term oxygen therapy or given indication for a Long-term oxygen therapy/ supplemental oxygen therapy for exercise
* Age: 18 to 80 years
* Participation in an inpatient pulmonary rehabilitation program (Schoen Klinik BGL, Germany)
* Written informed consent

Exclusion Criteria:

- Acute exacerbation of underlying pulmonary disease requiring cessation of exercise training.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | Day 1 to 5 and 6 to 10
  Change of dyspnea sensation rated by modified Borg scale (0 to 10) taken before and after exercise training

SECONDARY OUTCOMES:
Change of oxygen saturation (SpO2) during exercise training | Day 1 to 5 and 6 to 10
  SpO2 measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland).
Change of transcutaneous partial CO2 pressure (TcPCO2) during exercise training | Day 1 to 5 and 6 to 10
  TcPCO2 measured by continuous transcutaneous recording via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Change of heart rate during exercise training | Day 1 to 5 and 6 to 10
  Heart rate measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland).
Change of capillary partial pressure of CO2 (pCO2) during exercise training | Day 1 to 5 and 6 to 10
  pCO2 measured by capillary blood gases taken before and after the exercise training
Change of capillary partial pressure of O2 (pO2) during exercise training | Day 1 to 5 and 6 to 10
  pO2 measured by capillary blood gases taken before and after the exercise training
Change of inspiratory capacity (IC) during exercise training | Day 1 to 5 and 6 to 10
  IC measured by Spirometry taken before and after exercise training via SpiroSense Pro® (Pari, Starnberg, Germany)
Time to desaturation (SpO2 <=90%) and to severe desaturation (SpO2 <=85%) during exercise training | Day 1 to 5 and 6 to 10
  SpO2 measured by continuous transcutaneous recordung via Sentec-Digital Monitor® (Sentec, Therwil, Switzerland)
Assessment of leg fatigue via BORG scale | Day 1 to 5 and 6 to 10
  Change of leg fatigue assessed by modified Borg scale (0 to 10) taken before and after exercise training
Patients sensation regarding the oxygen delivery system | Day 5 and 10
  Patients will be asked to rate their experienced comfort after Session 1 and Session 2 via a 5-point Likert Skale: strongly agree, agree, neutral, disagree, strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Rembert Koczulla, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (1):
- Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee, Bavaria, Germany

REFERENCES:
- [Background] Kofod LM, Westerdahl E, Kristensen MT, Brocki BC, Ringbaek T, Hansen EF. Effect of Automated Oxygen Titration during Walking on Dyspnea and Endurance in Chronic Hypoxemic Patients with COPD: A Randomized Crossover Trial. J Clin Med. 2021 Oct 20;10(21):4820. doi: 10.3390/jcm10214820. PMID 34768338
- [Background] Schneeberger T, Jarosch I, Leitl D, Gloeckl R, Hitzl W, Dennis CJ, Geyer T, Criee CP, Koczulla AR, Kenn K. Automatic oxygen titration versus constant oxygen flow rates during walking in COPD: a randomised controlled, double-blind, crossover trial. Thorax. 2023 Apr;78(4):326-334. doi: 10.1136/thoraxjnl-2020-216509. Epub 2021 Oct 16. PMID 34656996
- [Background] Vivodtzev I, L'Her E, Vottero G, Yankoff C, Tamisier R, Maltais F, Lellouche F, Pepin JL. Automated O2 titration improves exercise capacity in patients with hypercapnic chronic obstructive pulmonary disease: a randomised controlled cross-over trial. Thorax. 2019 Mar;74(3):298-301. doi: 10.1136/thoraxjnl-2018-211967. Epub 2018 Aug 30. PMID 30166425